CLINICAL TRIAL: NCT05281419
Title: Combined Intralesional Triamcinolone Injection With Whole Breast Detection Radical Surgery in Treating Refractory Granulomatous Lobular Mastitis: A Randomized Controlled Trial
Brief Title: Combined Intralesional Triamcinolone Injection With Whole Breast Detection Radical Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Gaosong Wu, Ph D, MD, Chair, Department of Thyroid and Breast Surgery, Zhongnan Hospital of Wuhan University, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020091
Record Dates: First submitted 2022-01-07; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Refractory Granulomatous Lobular Mastitis
Keywords: Granulomatous lobular mastitis; Corticosteroids; Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intralesional triamcinolone injection with whole breast detection radical surgery (Experimental)
  Interventions: Other: Intralesional triamcinolone injection
- Whole breast detection radical surgery (Active Comparator)
  Interventions: Other: No intralesional triamcinolone injection

INTERVENTIONS:
Other: Intralesional triamcinolone injection — Injecting 40mg triamcinolone into the abscess cavity through the aspiration needle or drainage tube every 1 week
  Arms: Intralesional triamcinolone injection with whole breast detection radical surgery
Other: No intralesional triamcinolone injection — No intralesional triamcinolone injection
  Arms: Whole breast detection radical surgery

SUMMARY:
Granulomatous lobular mastitis (GLM) is a rare, chronic benign inflammatory disease of the breast, of unknown etiology. Pathologically, GLM typically manifests as non-caseating granulomatous lesions with leukomonocytes, lymphocytes, neutrophils and multinucleated giant cells, located in the center of breast lobules. With a rapidly increasing morbidity in the last two decades, GLM tends to occur in child-bearing women with a prolonged and recurrent course. Intralesional injection and topical corticosteroids can effectively reduce the side effects, especially in patients suffering from concomitant skin lesions (e.g., fistula, skin erosions, ulcers).For patients with diffuse disease, recurrence, or ineffective conservative treatment, wide local excision can be applied.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were pathologically diagnosed as refractory granulomatous lobular mastitis.
* Lesions are extensively distributed to more than three quadrants or with abscesses, sinus, fistula and persistent wound infection (skin ulceration and pus).
* Patients voluntarily participate in studies with informed consent.

Exclusion Criteria:

* History of breast surgery.
* Patients who choose conservative treatment.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recovery rate | Up to two years
  Disappearance of conscious symptoms: disappearance of pain and swelling sensations; disappearance of corresponding preoperative signs: clinically untouchable proto-inflammatory lesions, healing of wounds, ulcers, fistulas, sinus tracts, etc., no redness and rupture of the skin, no discharge of nipples, no inverted, no deformation, no upper and lower extremity nodular erythema and joint pain; recovery of imaging performance: no obvious hypoechondria under ultrasound, irregular masses without echo or mixed echoes, no preoperative dense punctate echoes, tubular echoes, abscesses or necrosis, liquefaction areas. Failure to meet the above criteria and maintain for more than one year without recurrence is defined as cure.
Recurrence rate | Up to one year
  Intraoperative inflammatory changes in the ipsilateral breast within one year of surgery, with lumps, abscesses, or fistula formation, with or without erythema nodosum of the upper and lower extremities and joint pain

SECONDARY OUTCOMES:
Scores of breast shape and cosmetic effect after surgery | Up to six months
  Standards of Harris
Degree of satisfaction | Up to one year
  The postoperative shape of breast, treatment time, postoperative pain and impact on life were divided into 5 grades, 1 point was the most serious, 5 points were no impact, the scores were added together to obtain the final score, and the satisfaction survey was conducted on patients every 3 months.
Healing of incision | Up to six months
  Defined as the time from the first day after surgery to the healing of the surgical incision, the wound surface is dry, no exudation, and no surgical incision complications occurs.
Complications of surgical incision | Up to one year
  Delayed incision healing, bleeding, hematoma, infection, fat liquefaction

CONTACTS AND LOCATIONS:
Locations (1):
- Qianqian Yuan, Wuhan, Hubei, China